CLINICAL TRIAL: NCT03896308
Title: Test-retest Reliability of the Chinese Version of the Verbal Learning Test and Selective Reminding Test Among People With Mild Cognitive Impairment
Brief Title: Reliability of Chinese Version of Verbal Learning Test and Selective Reminding Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Other Study IDs: YM108036E
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Mild Cognitive Impairment; Test-retest Reliability
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mild cognitive impairment (MCI) is distinguished from healthy aging by cognitive difficulties that are greater than expected for one's age and education. Amnestic mild cognitive impairment (aMCI) is a major sub-type of MCI with noticeable impairments in memory. Approximately 12% of aMCI will progress to AD per year. There are two test to evaluate the effects on memory, but both without Chinese version. This study is to know the test-retest reliability of the Chinese version of the Verbal learning test and Selective reminding test among people with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥50 years
2. Complained of memory impairment
3. Chinese Version Verbal Learning Test 10-minute delays ≤ 6 words
4. MMSE score≥24 and CDR score=0.5
5. Activities of daily living are intact
6. DSM-IV criteria for the diagnosis of dementia is not met

Exclusion Criteria:

1. Any significant neurologic disease other than suspected incipient Alzheimer's disease
2. Psychotic features, contraindication of exercise... which could lead to difficulty complying with the protocol

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild cognitive impairment (MCI) is distinguished from healthy aging by cognitive difficulties that are greater than expected for one's age and education. Amnestic mild cognitive impairment (aMCI) is a major sub-type of MCI with noticeable impairments in memory. Approximately 12% of aMCI will progress to AD per year. Guidelines for MCI recommended: controlling vascular risk factors and focusing on behavioral interventions.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-05-25 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-19 (Estimated)

PRIMARY OUTCOMES:
Chinese Version of Verbal Learning Test | Change from baseline at two week
Chinese Version of Selective Reminding Test | Change from baseline at two week

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan